CLINICAL TRIAL: NCT01888354
Title: Pilot Clinical Trial of ACTHar Gel 14 Days Subcutaneous (SQ) Versus ACTHar Gel Five Days SQ for the Treatment of MS Exacerbations
Brief Title: Pilot Clinical Trial of ACTHar Gel 14 Days Subcutaneous (SQ)Versus ACTHar Gel Five Days SQ for the Treatment of MS Exacerbations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Staley Brod, Staley A. Brod, MD, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-12-0210
Record Dates: First submitted 2013-05-16; First posted 2013-06-27 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Sclerosis (MS)
Keywords: MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acthar Gel 80 IU x 14 days (Experimental): Acthar Gel 80 IU SQ x 14 days
  Interventions: Drug: H.P. Acthar Gel (repository corticotropin injection)
- Acthar Gel 80 IU x 5 days (Experimental): Acthar Gel 80 IU SQ x 5 days
  Interventions: Drug: H.P. Acthar Gel (repository corticotropin injection)

INTERVENTIONS:
Drug: H.P. Acthar Gel (repository corticotropin injection) — Acthar Gel 80 IU
  Other Names: Acthar; Repository Corticotropin Injection; ACTH Gel

SUMMARY:
This pilot study is designed as a prospective cohort study to determine whether standard subcutaneous (SQ) Highly-Purified (HP) Acthar Gel 14 days is superior to SQ HP Acthar Gel 5 days in the treatment of relapses or attacks in multiple sclerosis (MS).

DETAILED DESCRIPTION:
Evaluations and treatment will be administered as an outpatient in the Neurology Clinic. Each subject will be seen for MS relapse or exacerbation in the Neurology Clinic during a routine or semi-emergent visit. Patients will be offered an FDA approved treatment (ACTHar Gel) for MS attacks under a standard 14 day SQ protocol (standard 14 day SQ protocol (80 IU x 14 days) or a 5 day SQ protocol - (5 day subcutaneous protocol (80 IU x 5 days). Both protocols are within package insert guidelines. The subjects will be evaluated for Extended Disability Status Scales (EDSS), a standardized measure of clinical status in MS and the initial visit and 28 days later (and 90 days later). We will compare the change in EDSS outcomes between day 0 and day 28 (day 90) to determine if the 14 days is superior to 5 day protocol may be clinically equivalent. Patients will also be evaluated for walking, upper extremity function (9 hole peg test), cognition and vision.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects with MS having a relapse (attack) or exacerbation of MS. Acute symptomatic exacerbation of MS present for > 24 hours and < 14 days at screening with new or worsening symptoms, and with signs referable to the symptoms in the absence of a fever or active infection.
2. Diagnosis of a relapsing forms of multiple sclerosis before randomization as determined by Poser or McDonald Criteria (standard MS diagnostic criteria).
3. Expanded disability status scale (EDDS) between 2 and 6.5, inclusive at entry.
4. Episodes include study neurologist or neuro-ophthalmologist diagnosed: acute optic neuritis, cerebellar, brainstem dysfunction, myelitis, focal cerebral, and/or definitive focal sensory dysfunction.
5. New objective clinical finding other than the sensory exacerbation or the bowel/bladder signs alone. Sensory deficits alone will not qualify except for optic neuritis.
6. Subjects may continue on their current immunomodulation therapy such as interferons, glatiramer acetate, gilenya or natalizumab.
7. Identified patients must be between the ages of 18 and 55 years, inclusive.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subjects who are pregnant, or nursing.
2. Any patients treated with systemic corticosteroid use within one month of the index episode at screening.
3. Prior use of immunosuppressive treatments within 90 days of index episode (mitoxantrone, azathioprine, Cellcept, IVIg) or plasmapheresis.
4. Unable to perform timed 25 foot walk (ambulation Index), 9 HPT (9 hole peg test), PASAT (Paced Auditory Serial Addition Test) 3.
5. Peripheral or cranial neuropathy as sole problem of acute episode.
6. Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
7. History of any significant cardiac, gastrointestinal, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude corticosteroid therapy.
8. Subjects with clinical diagnosis of scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of a peptic ulcer, congestive heart failure, hypertension, or sensitivity to proteins of porcine origin.
9. Primary Progressive Multiple Sclerosis (PPMS) (MS without attacks). -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comparison of EDSS Mean Recovery between 5-day vs 14-day SQ 80 IU ACTHar Gel therapy groups | 28 Days (with 90 day follow-up)
  To determine whether a standard 14 day course of SQ 80 IU ACTHar Gel therapy might be superior (in twice as many patients) to treatment with 5 day SQ regimen for ACTHar Gel as determined by EDSS mean recovery from Day 0 (time of steroid therapy initiation) to Day 28 (and day 90).

SECONDARY OUTCOMES:
Comparison of ambulation between the 5-day vs.14-day SQ 80 IU ACTHar Gel therapy groups | 28 Days (with 90 day follow-up)
  The ambulation index (AI) will be used for patients with long track (pyramidal) relapses, i.e. relapses with leg involvement. This is a standardized rating scale developed to assess mobility by evaluating the time and degree of assistance required to walk 25 feet.
Comparison of upper extremity function between the 5-day vs.14-day SQ 80 IU ACTHar Gel therapy groups | 28 day (with 90 follow up)
  The nine-hole peg test (9HPT) will be used for patients with arm involvement during relapses. The 9-HPT is a brief, standardized, quantitative test of upper extremity function. This is a timed test to determine how long it takes the patient to quickly place nine pegs (one at a time) in a wooden box with 9 empty holes, and them remove them again (one at a time) as quickly as possible. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand.
Comparison of subjective impressions of effectiveness between the 5-day vs 14-day SQ 80 IU ACTHar Gel therapy groups | 28 day (with 90 day follow up)
  The patient global impression of change (PGI-Change) will be used in patients to compare subjective impressions of effectiveness between treatment groups
Compare visual function between 5-day vs 14-day SQ 80 IU ACTHar Gel therapy groups | 28 day (with 90 day follow up)
  Visual function, as measured by low contrast Sloan sensitivity testing (LCSST) will be performed on each patient at baseline and at the end of treatment
Comparison of cognitive function between the 5-day vs 14-day SQ 80 IU ACTHar Gel therapy groups | 28 day (with 90 day follow up)
  In patients who report cognitive deficits during relapse, the paced auditory serial addition test (PASAT-3) will be used to assess and measure capacity and rate of information processing, and sustained and divided attention. This is a common neuropsychological test used in MS trials that involves working memory, attention and arithmetic capabilities. Patients will hear a series of recorded single-digit numbers at a rate of 1 per 3 seconds, and asked to add the number they just heard with the number they heard before.

OTHER OUTCOMES:
Comparison of MRI brain activity before and after ACTH treatment between the two treatment groups | 28 Days (with 90 day follow-up)
  Brain MRI scan ± Gd will be performed on subjects at entry, day 28 and day 90. Qualitative assessments of changes in numbers of Gd+ lesions from entry to exit will be assessed.
Comparison of immune changes before and after ACTH treatment between the two treatment groups | 28 Days (with 90 day follow-up)
  Peripheral mononuclear cells will be collected from patients at baseline,14 and 28 days post treatment and cytokine responses will be examined using a customized Human Cytokine Inflammatory Antibody Array including Th1-like (IL-2, IL-17, IFN-g, TNF-a, IL-1b), Th2-like cytokines (IL-4, IL-10, IL-13)

CONTACTS AND LOCATIONS:
Overall Officials: Staley A. Brod, MD, Principal Investigator — The Universtiy of Texas-Houston
Locations (2):
- United States (2):
  - The MS Center at the Neurology Center in Southern California, Oceanside, California
  - The University of Texas-Houston Neurology Clinic, Houston, Texas